CLINICAL TRIAL: NCT01253369
Title: A Phase II Study of Pazopanib in Patients With Relapsed or Refractory Small Cell Lung Cancer (SCLC)
Brief Title: Pazopanib in Patients With Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, David M. Jackman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-125; 113115 (Other: GlaxoSmithKline)
Record Dates: First submitted 2010-11-17; First posted 2010-12-03 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Small Cell Lung Cancer; Lung Cancer; SCLC
Keywords: pazopanib
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Pazopanib was given at a dose of 800 mg orally once per day for 28 day cycles (+/- 3 days). Patients received treatment as long as they were receiving clinical benefit.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient

SUMMARY:
Pazopanib is a drug that inhibits proteins thought to be important for new blood vessel formation. This drug has been used in other cancer research studies and information from those studies suggests that pazopanib may help block proteins that are important for the growth, invasion, and spread of cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

- To determine the progression-free survival rate in participants with relapsed or refractory small cell lung cancer who have received one prior regimen of systemic chemotherapy at 8 weeks

Secondary

* To determine the response rate (as measured by RECIST 1.1 criteria and changes in blood flow/perfusion as measured by perfusion CT)
* To determine median and overall survival
* To characterize the toxicity profile of pazopanib in this patient population.

Exploratory

* To analyze levels of circulating biomarkers from blood and urine samples obtained serially throughout the study and assess the utility of individual or subsets of these proteins to serve as a surrogate marker for treatment effect, treatment efficacy, and for tumor progression
* To measure and investigate the use of monocytes as surrogate markers of angiogenesis inhibition
* To analyze the subject population by identification of intra-tumoral biomarkers (such as c-kit, VEGF receptors, and microvessel density measured in available tumor biopsies) associated with the efficacy, safety and resistance to pazopanib
* To assess the utility of perfusion CT scan in evaluating changes in anti-angiogenic activity as a measure of treatment efficacy

STATISTICAL DESIGN: This study uses a two-stage design to evaluate efficacy of cetuximab based on progression-free rate (PFR) at week 8 defined as complete response (CR), partial response (PR) or stable disease (SD) per RECIST 1.1 criteria. The null and alternative PFR are 30% and 50%. If fewer than 4 patients enrolled in the stage one cohort (n=15 patients) achieve SD or better than accrual would not proceed to stage two (n=15 patients). If 13 or more patients are progression-free of the 30 patients then the null hypothesis will be rejected. The probability that the treatment will be considered promising if the true PFR rate was 30% is 8.4% and 82% if the true PFR rate was 50%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of small cell neuroendocrine carcinoma based on either histology or cytology with radiologically-confirmed progressive disease.
* Participants should have received first-line chemotherapy and may have had up to two prior chemotherapy regimens. Radiation therapy may have been part of the permitted prior therapy.
* Participants with brain metastases will be allowed if they have been treated with surgery and/or radiation therapy more than 21 days prior, are asymptomatic, and are stable for at least one week off steroids.
* 18 years of age or older
* ECOG Performance status of 0, 1 or 2
* Ability to swallow and retain oral medication
* Disease must be measurable according to RECIST 1.1
* Adequate organ function as defined in the protocol

Exclusion Criteria:

* Prior malignancy except for participants that have been disease-free for 3 years or with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma
* History or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for one week prior to first dose of study drug.
* Clinically significant gastrointestinal abnormalities
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480msecs
* History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting; myocardial infarction; unstable angina; symptomatic peripheral vascular disease; Class III or IV congestive heart failure
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism or insufficiently treated deep venous thrombosis within the past 6 months
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture or ulcer
* Evidence of active bleeding or bleeding diathesis
* Hemoptysis in excess of 2.5mL within 6 weeks of first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Use of any prohibited medication within the timeframes listed in the protocol
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug
* Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors
* Is now undergoing and/or has undergone in the 14 days immediately prior to first dose of study drug, any cancer therapy
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jackman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Gandhi L; Heist RS; Lucca JV; Temel JS; Fidias P; Morse LK; Johnson BE; Dana-Farber Cancer Institute, Boston, MA; Massachusetts General Hospital Cancer Center, Boston, MA. A phase II trial of pazopanib in relapsed/refractory small cell lung cancer (SCLC). J Clin Oncol 2012; 30 (suppl; abstr 7099)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from November 2010 through April 2012.
Period: Overall Study
Arm/Group | Pazopanib
Started | 33
Evaluable | 30 (Evaluable pts were w/ measurable disease, min 1 cycle of trt rcvd and 1 on-trt disease assessment.)
Completed | 0 (Since treatment duration was not fixed, patients were not considered to have completed treatment.)
Not Completed | 33
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Progressive disease | 23
Not completed — Not Evaluable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 61 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 33
Response to 1st Line Therapy [Number; unit: participants]
  Chemo-Refractory | 18
  Chemo-Sensitive | 15

OUTCOME MEASURES:

1. Primary Outcome: 8-Week Progression-Free Rate
Description: The 8-week progression free rate (PFR) was defined as achieving complete response (CR), partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria by the time of the first disease assessment (8 weeks). Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions; PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD; and SD is neither sufficient decrease to qualify as PR nor sufficient increase to qualify as progressive disease (PD). PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. Response needed confirmation within 4 weeks. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions.
Time Frame: For this endpoint, disease was evaluated radiologically at baseline and week 8 on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 3 cycles range (1-20).
Population: The analysis dataset is comprised of evaluable patients. Patients who had measurable disease at baseline, received at least 1 cycle of therapy and had their disease re-evaluated were considered evaluable for response.
Measure: Number (80% Confidence Interval); unit: proportion of patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 30
proportion of patients | 0.567 [0.434 to 0.692]

2. Secondary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better objective response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 3 cycles range (1-20).
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: proportion of patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 30
proportion of patients | 0.033 [0.004 to 0.124]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv4.
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 12/33
Other Adverse Events (participants affected / at risk) | 26/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=33)
Cardiac disorders - Other, specify (Cardiac disorders) | 4
Heart failure (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lipase increased (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Memory impairment (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=33)
Anemia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5
Cardiac disorders - Other, specify (Cardiac disorders) | 6
Supraventricular tachycardia (Cardiac disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 10
Pancreatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Edema face (General disorders) | 1
Fatigue (General disorders) | 13
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 8
Bruising (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 2
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 2
Weight loss (Investigations) | 5
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Nervous system disorders - Other, specify (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No